CLINICAL TRIAL: NCT03846687
Title: Validation of the Modified Foot Function Index (mFFI) for Use in Hallux Valgus
Brief Title: Validation of Patient Reported Outcome Measures for Use in Hallux Valgus
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: D-FR-52120-257
Record Dates: First submitted 2019-02-13; First posted 2019-02-20 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Hallux Valgus
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to explore whether the mFFI is fit for purpose in adults with hallux valgus (HV).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, of any race and, aged ≥ 18 years
* Clinical diagnosis of hallux valgus
* Fluent in reading/speaking US-English to read and understand informed consent form and to participate in the interview

Exclusion Criteria:

* Participation in another foot-based clinical trial in the last 90 days or in Ipsen's clinical trial D-FR-52120-237
* Current chronic drug or alcohol abuse problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects referred by clinicians
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Concept elicitation (CE) of mFFI | 7 days
  Face-to-face interview (approx. 25 minutes), using semi-structured interview guide to explore the symptoms and impact of HV.
Cognitive debriefing (CD) of mFFI | 7 days
  Face-to-face interview (approx. 25 minutes) to explore understanding and relevance of mFFI items.
Usability testing of mFFI | 7 days
  Telephone interview (approx. 20 minutes) using a semi-structured interview guide to explore how participants found usability of completing the mFFI daily in electronic format on their own device.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (3):
- United States (3):
  - University Foot and Ankle Institute, Santa Monica, California
  - Ankle and Foot Care Centers, Youngstown, Ohio
  - Futuro Clinical Trials, LLC, McAllen, Texas